CLINICAL TRIAL: NCT03080779
Title: The Incidence of Chronic Headache and Low Back Pain After Accidental Dural Puncture (ADP) With a Tuohy Needle and Epidural Blood Patch in the Obstetric Population: A Prospective 2-group Cohort Multicentre Study
Brief Title: Long Term Outcomes After Accidental Dural Puncture ADP Study
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: UHLeicester
Record Dates: First submitted 2016-12-20; First posted 2017-03-15 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Post-Dural Puncture Headache; Chronic Headache; Chronic Low Back Pain
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADP Group: Index group includes participants who have suffered an accidental dural puncture with a 16 gauge Tuohy needle
- Non-ADP group: Control group includes participants who received an uneventful epidural analgesia with a 16 gauge Tuohy needle

SUMMARY:
Post Dural Puncture Headache (PDPH) causes significant short-term disability, prevents mobilisation, affects childcare activities and results in prolonged hospital stay. Initial treatment involves painkillers and if patient fails to respond, an Epidural Blood Patch (EBP). EBP involves taking patient's blood and injecting into the epidural space. It is generally agreed that PDPH is a self-limiting condition and resolves in two weeks. However there is emerging evidence that patients with PDPH could be at an increased risk of developing longstanding (chronic) headaches. Retrospective case studies show that between 28 - 34% of patients who developed PDPH had longstanding headaches at 18 months after the insertion of the epidural. There is also recent evidence of new onset low back pain developing in patients who have received an epidural blood patch that was performed to treat PDPH. Nearly two thirds of patients from a hospital in UK had new onset low back pain after they had received epidural blood patch treatment. Presently, there is no prospective clinical study evaluating the development of longstanding headaches and new onset low back pain after the development of PDPH. Aim of the present study is to evaluate the incidence of longstanding headache after accidental dural (ADP) puncture and the incidence of new onset low back pain after epidural blood patch treatment.

DETAILED DESCRIPTION:
Headache can be a complication after insertion of an epidural needle for pain relief during labour. The headache is called Post Dural Puncture Headache (PDPH). PDPH causes significant short-term disability, prevents mobilisation, affects childcare activities and results in prolonged hospital stay. Initial treatment involves painkillers and if patient fails to respond, an Epidural Blood Patch (EBP). EBP involves taking patient's blood and injecting into the epidural space. It is generally agreed that PDPH is a self-limiting condition and resolves in two weeks. However there is emerging evidence that patients with PDPH could be at an increased risk of developing longstanding (chronic) headaches. Retrospective case studies show that between 28 - 34% of patients who developed PDPH had longstanding headaches at 18 months after the insertion of the epidural. There is also recent evidence of new onset low back pain developing in patients who have received an epidural blood patch that was performed to treat PDPH. Nearly two thirds of patients from a hospital in UK had new onset low back pain after they had received epidural blood patch treatment. Presently, there is no prospective clinical study evaluating the development of longstanding headaches and new onset low back pain after the development of PDPH.

Aim of the present study is to evaluate the incidence of longstanding headache after accidental dural (ADP) puncture and the incidence of new onset low back pain after epidural blood patch treatment.

Methods: The proposed study is a prospective, cohort study that will be conducted at six centres (Leicester, Derby, Bradford, Colchester, Bedford and Cambridge) over 36 months. Index participants who suffer ADP will be matched with control participants who have received an uneventful epidural insertion. The index and control participants will be matched for age, body weight, parity and the type of delivery. Mothers who have longstanding headache or low back pain will be excluded form the study. After providing written consent, the participants will be provided with a questionnaire pack containing three sets of two questionnaires to be completed at 6, 12 and 18 months after developing the headache as well as stamped envelopes to return the questionnaires to the research team. A research team member will perform telephone follow up 6, 12 and 18 months to encourage completion of the questionnaires. Participation in the study will end at 18 months after completion of the study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Index: Participants aged over 18 years who have sustained accidental dural puncture with 16-gauge Tuohy needle
* Control: Participants aged over 18 years who have received uneventful epidural insertion with 16-gauge Tuohy needle

Exclusion Criteria:

* Lack of consent including from those participants who lack mental capacity to give informed consent
* Pre-existing chronic headache (the patients suffer from 15 or more headache days every month)
* Pre-existing chronic low back pain (the patients suffer from 7 or more low back pain days every month)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obstetric
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-06-27 (Actual)

PRIMARY OUTCOMES:
The incidence of chronic headache at 18 months in the ADP group when compared to the control non-ADP group | 18 months
  Questionnaire

SECONDARY OUTCOMES:
The incidence of chronic low back pain at 18 months in the ADP group when compared to the control non-ADP group. | 18 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: N Gopinath, Principal Investigator — University Hospitals, Leicester
Locations (3):
- United Kingdom (3):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Bedford Hospitals NHS Trust, Bedford
  - Royal Derby Hospitals, Derby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niraj G, Mushambi M, Gauthama P, Patil A, Kelkar A, Hart E, Nurmikko T; Accidental Dural Puncture Outcome Study Collaborative Group. Persistent headache and low back pain after accidental dural puncture in the obstetric population: a prospective, observational, multicentre cohort study. Anaesthesia. 2021 Aug;76(8):1068-1076. doi: 10.1111/anae.15491. Epub 2021 Apr 23. PMID 33891312